CLINICAL TRIAL: NCT07382115
Title: Clinical and Radiographic Comparison of Indirect Pulp Treatment and Direct Pulp Capping in Deep Carious Primary Second Molars: One-Year Results
Brief Title: Indirect and Direct Pulp Therapy in Primary Second Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ozlem Beren SATILMIS, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/07
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Deep Dentin Caries in Primary Teeth; Pulp Therapy in Primary Molars
Keywords: indirect pulp treatment; direct pulp capping; Mineral trioxide aggregate; Randomized controlled trial; Primary second molars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect Pulp Treatment (IPT) (Experimental): Teeth allocated to this arm received indirect pulp treatment. Selective caries removal was performed, leaving affected dentin over the pulp, followed by placement of mineral trioxide aggregate (MTA) and restoration with a stainless steel crown (SSC).
  Interventions: Procedure: Indirect Pulp Treatment
- Direct Pulp Capping (DPC) (Experimental): Teeth allocated to this arm received direct pulp capping. After <1 mm pulp exposure, mineral trioxide aggregate (MTA) was placed directly over the exposed pulp tissue, followed by restoration with a stainless steel crown (SSC).
  Interventions: Procedure: Direct Pulp Capping

INTERVENTIONS:
Procedure: Indirect Pulp Treatment — Selective caries removal was performed, leaving affected dentin over the pulp. Mineral trioxide aggregate (MTA) was placed, followed by restoration with a stainless steel crown (SSC).
  Arms: Indirect Pulp Treatment (IPT)
Procedure: Direct Pulp Capping — After <1 mm pulp exposure, mineral trioxide aggregate (MTA) was placed directly over the exposed pulp tissue, followed by restoration with a stainless steel crown (SSC).
  Arms: Direct Pulp Capping (DPC)

SUMMARY:
The purpose of this randomized controlled clinical trial was to compare the clinical and radiographic outcomes of indirect pulp treatment (IPT) and direct pulp capping (DPC) using mineral trioxide aggregate (MTA) in deep carious primary molars. Children with deep dentin caries in primary molars were randomly assigned to receive either IPT or DPC. Clinical and radiographic evaluations were performed at 6 and 12 months to assess treatment success. The findings of this study aim to provide evidence-based guidance for the management of deep dentin caries in primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy children aged 7 to 9 years
* Primary second molars with deep dentin caries indicated for vital pulp therapy
* Absence of clinical signs or symptoms of irreversible pulpitis
* No spontaneous or prolonged pain
* Teeth with no tenderness to percussion or palpation
* No pathological mobility, swelling, fistula, or abscess
* Radiographic findings showing intact lamina dura and normal periodontal ligament space
* Absence of periapical or furcation radiolucency
* No evidence of pathological internal or external root resorption
* Teeth considered restorable
* Written informed consent obtained from parents

Exclusion Criteria:

* Children with systemic diseases or medical conditions affecting healing
* Teeth with signs or symptoms of irreversible pulpitis
* Presence of spontaneous pain, night pain, or prolonged pain
* Teeth with periapical or furcation radiolucency
* Teeth with pathological internal or external root resorption
* Presence of pulpal calcifications or pulp stones
* Non-restorable teeth
* Lack of parental consent

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Clinical success of indirect pulp treatment and direct pulp capping | 12 months
  Clinical success was defined as the absence of spontaneous pain, swelling, fistula, pathological mobility, or tenderness to percussion.
Radiographic success of indirect pulp treatment and direct pulp capping | 12 months
  Radiographic success was defined as the absence of periapical radiolucency, internal or external root resorption, pathological changes, or other radiographic signs of pulpal or periapical pathology during the follow-up period.

SECONDARY OUTCOMES:
Effect of pulp exposure location on treatment success | 12 months
  The location of pulp exposure (occlusal or proximal) was recorded and its association with clinical and radiographic success of vital pulp therapy was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No